CLINICAL TRIAL: NCT01119248
Title: Pediatric Temperature Variation in the MRI Scanner Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Anuradha Patel, Associate Professor, Dept. of Anesthesiology, Rutgers, The State University of New Jersey
Other Study IDs: 0120100053
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Children Requiring MRI
Keywords: Children MRI General Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children undergoing MRI: 120 children ages of 6 months and 8 years for MRI and axillary temperature before MRI and after the MRI with MRI compatible device
  Interventions: Other: axillary temperature before MRI and after the MRI

INTERVENTIONS:
Other: axillary temperature before MRI and after the MRI — observation of body temperature changes with axillary temperature measurement with MRI compatible device

SUMMARY:
The number of children undergoing MRI imaging has increased significantly in the past years, because many young children cannot stay still for the duration of the scan, have difficulty tolerating the confined space and the noise produced by the Magnetic Resonance Imaging (MRI) machine, sedation or General Anesthesia is required in these cases. In the investigators institution, the investigators use General Anesthesia for children undergoing MRI.

Because children have a larger surface area to body weight ratio; hypothermia from passive heat loss is one of the anesthesiologists' concerns.

MRI requires a cool environment with low humidity; this specialized environment represents a significant thermal challenge to the anesthetized children. Since most temperature devices are not compatible with the MRI, the simple task to measure temperature change has never been investigated.

DETAILED DESCRIPTION:
It is known that following the induction of anesthesia, core hypothermia occurs in three stages;

1. Redistribution
2. Linear phase
3. Plateau phase Redistribution This accounts for the largest drop in core temperature of the three stages. Vasodilatation causes redistribution of heat from the core to the periphery.

Linear Phase This begins at the start of surgery as the patient is exposed to cold cleaning fluids and cool air flow in the theatre. Heat loss exceeds heat production, and most surgery does not extend past the linear phase.

* Radiation contributes the most (40%) and is proportional to environment/core, temperature difference to the power of four.
* Convection contributes up to 30% and is proportional to air velocity.
* Conduction contributes up to 5% and is proportional to the difference in surface temperatures.
* Evaporation contributes up to 15% and occurs from cleaning fluids, skin, respiratory and wound. A laparotomy can contribute up to 50% of the total.
* Respiratory contributes 10% (8% evaporation of water; 2% heating of air) and is enhanced by the cooling effect of cold anesthetic gases.
* Cold intravenous fluids. Plateau Phase Once core temperature falls below the thermoregulatory threshold, peripheral vasoconstriction increases and acts to limit the heat loss from the core department. When core heat production = heat loss to the peripheral compartment, core temperature reaches a plateau. Patients with an autonomic neuropathy (diabetics) have impaired sympathetic vasoconstriction and are unable to establish a core plateau in phase 3. Combined general and regional anesthesia will have a similar effect as the regional anesthetic (spinal/epidural) will prevent vasoconstriction in the legs; i.e. failure to establish a core plateau.

The ability to maintain body temperature is also compromised because anesthesia impairs intrinsic thermoregulatory response.

Heating devices including fluid warmers and bear huggers, commonly used in the Operating Room theaters, are incompatible with MRI.

On the other hand, MRI produces Radiofrequency Energy that transforms into heat within the patient's tissues. This may partially offset the heat loss.

The purpose of our study is to determine if children undergoing MRI under General Anesthesia become hypothermic and whether aggressive measures should be taken to prevent passive heat loss during MRI studies.

Study Design This is an observational, prospective non blinded study.

ELIGIBILITY:
Inclusion Criteria:

* 6 months to 8 years undergoing general anesthesia for elective MRI of brain, spine and extremities. Patients who were ASA physical status 1-3 only were included.

exclusion criteria: Patients who were ASA 4-5 were excluded from the study. Patients not NPO for solids for 8 hours and liquids for 2 hours were excluded.

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 6 months to 8 years
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Patel, MD, Principal Investigator — Rutgers-NJMS
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in radiology department in MRI holding area.
Groups:
- Children Undergoing MRI: children ages 6 months to 8 years scheduled for MRI under general anesthesia
Period: Overall Study
Arm/Group | Children Undergoing MRI
Started | 120
Completed | 115
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Population: children scheduled for MRI under general anesthesia
Groups:
- Not Applicable: prospective observational cohort study
Arm/Group | Not Applicable
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 120
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 63
Region of Enrollment [Number; unit: participants]
  United States | 120
Body Surface Area (BSA) [Mean (Full Range); unit: m²] | 0.68 [0.29 to 1.40]

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Temperature in Children Undergoing MRI Under General Anesthesia (GA)and Change in Room Temperature Before and After MRI
Description: Axillary temperature was measured with MRI-compatible Tempa dot immediately before general anesthesia was induced. Second axillary temperature reading was taken at the conclusion of the MRI scan before emergence from general anesthesia. Room temperature was measured with a digital thermometer placed in scanner room outside the magnet range.
Time Frame: prior to induction of general anesthesia and at conclusion of MRI an average of two hours
Population: 120 children were enrolled for the prospective cohort study. 5 children were excluded from the study: 3 did not fit study criteria after enrollment before start of the procedure, one did not get any intravenous fluids during scan, the MRI scan was cancelled after enrollment in one patient
Measure: Mean (Full Range); unit: celsius degrees
Groups:
- Children Undergoing MRI: children 6 months to 8 years requiring GA for MRI
Arm/Group | Children Undergoing MRI
Number analyzed (Participants) | 115
celsius degrees
  preMRI temperature | 36.7 [35.7 to 37.7]
  post MRI temperature | 36.3 [34.3 to 38.1]
  difference in body temperature | -0.4 [-2.9 to 1.6]
  Pre MRI room temperature | 21.1 [16.1 to 25.6]
  post MRI room temperature | 21.3 [16.1 to 25.6]
  Difference in Room temperature | 0.2 [0.1 to 0.3]
Statistical Analysis 1: Comparison: Children Undergoing MRI; Test type: Superiority or Other; p < .001, t-test, 2 sided; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.48 to -0.25], Standard Deviation 0.62

2. Secondary Outcome: Relationship Between Pre MRI Body Temperature and Change in Body Temperature After MRI
Description: Bivariate analysis between pre MRI body temperature and change in body temperature after MRI. Body temperature of the subjects was measured with MRI compatible Tempadot. Reported is the change in body temperature after MRI with 1 degree increase in body temperature between subjects after adjusting for body surface area (BSA), type of MRI and duration of MRI. A positive change value reflects a child who was 1 degree C warmer experienced greater warming. The negative change reflects that a child who was 1 degree C warmer experienced greater cooling.
Time Frame: Prior to start of general anesthesia and immediately after completion of MRI an average of two hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: celsius degrees
Arm/Group | Children Undergoing MRI
Number analyzed (Participants) | 115
celsius degrees | -0.69 [-0.95 to -0.43]
Statistical Analysis 1: Comparison: Children Undergoing MRI; pre- MRI body temperature was associated with change in body temperature after MRI by bivariate analysis. The values presented are adjusted for body surface area, type of MRI, room temperature and duration of MRI; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-0.95 to -0.43]

3. Secondary Outcome: Relationship Between Body Surface Area (BSA) and Change in Body Temperature After MRI
Description: Bivariate analysis between BSA and change in body temperature after MRI. Reported is the change in body temperature after MRI with 1m2 increase in BSA, after adjusting type of MRI and duration of MRI. A positive change value reflects increase in body temperature with an increase in BSA and vice versa
Time Frame: Prior to start of general anesthesia and immediately after completion of MRI scan an average of two hours
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: celsius degrees
Arm/Group | Children Undergoing MRI
Number analyzed (Participants) | 115
celsius degrees | .52 [.23 to .82]
Statistical Analysis 1: Comparison: Children Undergoing MRI; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: until subject had fully recovered from anesthesia and was ready for discharge up to 2 hours
Groups:
- Children Undergoing MRI: infants 6 months to children 8 years
Arm/Group | Children Undergoing MRI
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

LIMITATIONS AND CAVEATS:
There was difficulty in collecting data due to the restricted MRI environment. We used Tempadot which is not a digital or electronic temperature measurement device and is MRI compatible, but the device may not be as accurate as the other devices

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes